CLINICAL TRIAL: NCT04337151
Title: Blood Titanium Analysis of Patients With MAGEC Spine Rods in the COVID-19 Environment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal National Orthopaedic Hospital NHS Trust (Other)
Responsible Party: Principal Investigator, Dr Harry Hothi, Implant Science Fellow, Royal National Orthopaedic Hospital NHS Trust
Other Study IDs: RNOH MAGEC
Record Dates: First submitted 2020-04-03; First posted 2020-04-07 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: MAGEC Rod

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: MAGEC Spine Rod — Magnetically controlled growing spine rod used for the surgical treatment of scoliosis.
Diagnostic Test: Titanium blood test — A blood test captured to measure the level of titanium

SUMMARY:
Magnetic Expansion Control (MAGEC) growth rods are used in the surgical treatment of children with scoliosis; the primary constituent metal alloy in these is titanium.

Since June 2019, the manufacturer has released two Urgent Field Safety Notices (FSN) relating to known issues with the function of the rods that increase the risk of early failure and unplanned revisions. The UK MHRA has issued two similar Medical Device Alerts (MDA) with the most recent MDA issued on 1st April 2020, stating that (1) MAGEC rods must not be implanted in the UK until further notice and (2) all patients already implanted with this device should be followed up as soon as is possible.

At the time of writing, hospitals across the world are facing incredible challenges in dealing with the COVID-19 pandemic. Due to this, virtually all planned clinic visits for MAGEC rod patients and X-ray appointments have been postponed to help reduce the risk of the virus spreading.

Recent retrieval studies have shown that mechanical wear and corrosion of these rods is common, with a risk that the debris generated is released into surrounding tissue. This wear and corrosion is thought to be the primary cause of implant failures and the underlying implant factors leading to the issuing of FSNs and MDAs.

Whilst titanium is known to be highly biocompatible, the baseline and toxic levels of this alloy in biological fluids are poorly understood. Additionally, a better understanding of blood titanium levels in patients with MAGEC rods may enable this to become a biomarker of wear and corrosion of the rods. This may help surgeons identify earlier those patients who may develop implant related problems.

Furthermore, in the current COVID-19 environment, a blood test to measure titanium levels may be one of the most suitable ways in which to continue patient monitoring (and identify those at greatest risk of implant related issues), in the absence of regular clinic visits.

Previous work from the RNOH involved a similar study investigating patients with titanium hip implants.

ELIGIBILITY:
Inclusion Criteria:

* Patients that have been treated with, and still have, a MAGEC rod.

Exclusion Criteria:

* Patients that do not have a MAGEC rod implant.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children being treated for early onset scoliosis.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-04 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Titanium level | Within 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Royal National Orthopaedic Hospital, Stanmore, United Kingdom

IPD SHARING:
Plan to Share IPD: No